CLINICAL TRIAL: NCT06421675
Title: A Study of Elranatamab Management With Outpatient and Intermittent Dosing in Relapsed/Refractory Multiple Myeloma
Brief Title: Outpatient and Intermittent Dosing of Elranatamab in Relapsed/Refractory Multiple Myeloma
Acronym: EMBRACE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Pfizer (Industry); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2023-EMBRACE
Record Dates: First submitted 2024-03-11; First posted 2024-05-20 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Refractory Multiple Myeloma
Keywords: relapsed; refractory; multiple myeloma; elranatamab; cytokine release syndrome; immune effector-cell associated neurotoxicity
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Cytokine Release Syndrome

STUDY DESIGN:
Intervention Model Description: Multi-center, single-arm, phase II study of single-agent elranatamab in patients with relapsed and/or refractory multiple myeloma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elranatamab injection (Experimental): The administration of two step-up elranatamab doses (12 mg and 32 mg) and full dose 76 mg. The dosing interval for the first Cycle (each cycle q28 days) is every week. Cycles 2-3, the dosing interval increases to q2weeks. Cycles 4-12, the dosing interval increases to q4weeks. Cycles 13+, further dosing interval increases to q8weeks will be scheduled if a participant meets criteria for IMWG complete response (CR) in Cycle 12 (bone marrow required at Cycle 12 to confirm). If a participant does not meet CR criteria at Cycle 12, they will be continued on Q4W dosing.
  Interventions: Drug: Elranatamab injection

INTERVENTIONS:
Drug: Elranatamab injection — Elranatamab (Elrexfio) is a humanized bispecific antibody that targets both BCMA-expressing multiple myeloma (MM) cells and CD3-expressing T cells.
  Other Names: Elrexio

SUMMARY:
A phase II study of single agent elranatamab in patients with relapsed and/or refractory multiple myeloma (MM) who have previously received at least three classes of therapeutic agents and are refractory to the last line of treatment. The primary objective of this study is to improve the tolerability and safety of elranatamab in patients with relapsed and/or refractory multiple myeloma by evaluating an outpatient and intermittent dosing strategy.

DETAILED DESCRIPTION:
This is a multi-centre, single arm, phase II study of single agent elranatamab in patients with relapsed and/or refractory multiple myeloma (MM) who have previously received at least three classes of therapeutic agents and are refractory to the last line of treatment. Potential study participants must have documented evidence of refractory or progressive disease during or within 60 days (measured from the end of the last cycle) of completing treatment with the last anti-myeloma drug regimen used just prior to study entry. Study participants will receive SC administration of elranatamab until disease progression, unacceptable toxicity or death. The primary short term outcome is hospitalization rate within the first 2 weeks of Cycle 1 of treatment; the primary long term outcome is rate of grade 3+ infections within the first 24 months of treatment. Study participants will be followed for survival for 36 months from the date of enrollment. A total of 40 study participants will be enrolled across approximately 5 Canadian clinical trial sites.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed and/or refractory MM defined as:

   1. Documented evidence of progressive disease (PD) after achieving at least minimal response (MR) for ≥ 1 cycle during a previous MM treatment (i.e., relapsed MM).
   2. Disease progression during or within 60 days from the end of the most recent MM treatment (i.e., refractory MM).
2. Measurable disease based on IMWG criteria, defined as at least one of the following, documented within 28 days before enrollment:

   1. Serum M-protein ≥ 0.5 g/dl.
   2. Urine M-protein excretion ≥ 200 mg/24 h.
   3. Serum-free light chains (FLC) assay: Involved FLC level ≥ 10 mg/dl (≥ 100 mg/l) AND an abnormal serum-free light chain ratio (< 0.26 or > 1.65) only for patients without measurable serum or urine M protein.
3. Receipt of at least three prior classes of drugs either in separate regimens or as combinations.

   The three classes are defined as:

   An immunomodulatory drug (lenalidomide or pomalidomide), a proteasome inhibitor (bortezomib, ixazomib, carfilzomib), and an anti-CD38 drug (daratumumab or isatuximab).
4. At least 18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2.

Exclusion Criteria:

Medical conditions

1. Active plasma cell leukemia (either 20% of peripheral white blood cells or > 2.0 × 109/L circulating plasma cells by standard differential).
2. Amyloidosis.
3. POEMS syndrome (Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal plasma cell disorder, Skin Changes).
4. Monoclonal gammopathy of unknown significance or smoldering multiple myeloma.
5. Solitary plasmacytoma.
6. Stem cell transplant within 12 weeks prior to enrollment or active graft versus host disease.
7. History of prior treatment with a BCMA targeting agent.

   Laboratory Parameters
8. Laboratory results within 28 days as per below prior to enrollment:

   * Absolute neutrophil count (ANC) ≤ 1.0 x 109 /L) (use of growth factor is permitted if completed at least 7 days prior to enrollment).
   * Platelet count ≤ 25 x 109 /L (transfusion support permitted if completed at least 7 days prior to enrollment).
   * Hemoglobin ≤ 8.0 g/dL (transfusion support permitted if completed at least 7 days prior to enrollment, concurrent erythropoietin stimulating agents allowed).
   * Serum AST and ALT > 2.5 x upper limit of normal (ULN).
   * Creatinine clearance < 30 mL/min (according to the Cockcroft Gault formula, by 24-hour urine collection for creatinine clearance, or according to local institutional standard method).
   * Total bilirubin > 2.0 x ULN (≥ 3.0 unless known to have Gilbert's disease).

   Support Requirement
9. As this protocol requires outpatient administration, the patient will be excluded if they cannot agree to the following for the first 9 days post-first dose of drug administration:

   1. Staying within 60 minutes of travel distance to their trial-based hospital.
   2. Must have a caregiver/support person who will stay with the patient.
   3. Patient and/or their caregiver/support person agree to monitor and record oral temperature q8 hours.
   4. Patients must agree that if they have an oral temperature of (≥38°C), they must report to the study team within 1 hour and can come to the hospital for admission within 2 hours.

   Other co-morbidities
10. Impaired cardiovascular function or clinically significant cardiovascular diseases, defined as any of the following within 6 months before enrollment:

    * Acute myocardial infarction or acute coronary syndromes (eg, unstable angina, coronary artery bypass graft, coronary angioplasty or stenting, symptomatic pericardial effusion).
    * Clinically significant cardiac arrhythmias (eg, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia).
    * Thromboembolic or cerebrovascular events (eg, transient ischemic attack, cerebrovascular accident, deep vein thrombosis [unless associated with a central venous access complication], or pulmonary embolism).
    * Prolonged QT syndrome (or triplicate average QTcF >470 msec at screening).
11. Ongoing Grade ≥2 peripheral sensory or motor neuropathy.
12. History of Guillain-Barre Syndrome (GBS) or GBS variants, or history of any Grade ≥3 peripheral motor polyneuropathy.
13. Unresolved acute effects of any prior therapy for MM in the last three months to either baseline severity or NCI CTCAE ≤Grade 1.
14. Active HBV, HCV, SARS-CoV2, HIV, or any active, uncontrolled bacterial, fungal, or viral infection.
15. Any other active malignancy within 2 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
16. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities), or surgical (major surgery within 14 days prior to enrollment) that could interfere with the patient's safety, obtaining informed consent or compliance to the study procedures.
17. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to elranatamab or any of the components of the study treatment.

    Concomitant Medications
18. Treatment with a chemotherapeutic or anti-MM drug within the last 28 days or 5 half-lives (whichever is shorter) prior to enrollment or are currently enrolled in another interventional clinical study.
19. Receipt of any other therapy to treat cancer (including radiation, biologics, cellular therapies, and/or steroids at doses > 20 mg dexamethasone or equivalent) within 14 days prior to the enrollment.
20. Receipt of any live vaccine within 30 days prior to enrollment or expected need of live vaccination during study participation. (Administration of locally approved non-live vaccine can be done as per local guidelines during the screening and/or treatment period including the COVID-19 mRNA vaccine. Elranatamab should be administered ± 7 days from the SARS-CoV-2 vaccine administration).

    Pregnancy and Contraception
21. Pregnancy or lactating female or inability of female patients of childbearing potential (FCBP) to meet contraception requirements (see Section 5.1.3.).

    Informed Consent
22. Inability to provide signed, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate | 2 weeks
  Hospitalization rate, defined as the number of patients who are hospitalized within the first 2 weeks of Cycle 1 of treatment, due to any cause, divided by the number of patients who are treated with elranatamab.
Rate of grade 3+ infections | 24 months
  Rate of grade 3+ infections as grade by NCI CTCAE v5 within the first 24 months of treatment, defined as the number of patients who experience a grade 3+ infection within 24 months of treatment, divided by the number of patients who are treated with elranatamab.

SECONDARY OUTCOMES:
Overall response rate. | 36 months
  Overall response rate, defined by the IMWG criteria.
Progression free survival. | 36 months
  PFS, defined as the time from the date of first dose until confirmed PD per IMWG criteria or death due to any cause, whichever occurs first.
Duration of response. | 36 months
  DOR is defined, for participants with an overall response per IMWG criteria, as the time from the first documentation of overall response that is subsequently confirmed, until confirmed PD per IMWG criteria, or death due to any cause, whichever occurs first.
Time to response. | 36 months
  TTR is defined, for participants with an overall response per IMWG criteria, as the time from the date of first dose to the first documentation of overall response that is subsequently confirmed.
Adverse Events | 36 months
  AEs will be graded according to NCI CTCAE Version 5. CRS and ICANS will be assessed. AEs will be characterized by type, frequency, severity, timing, seriousness, and relationship to elranatamab. AEs will be presented with and without regard to causality based on the investigator's judgment. The frequency of overall toxicity, categorized by toxicity Grades 1 through 5, will be described. Additional summaries will be provided for AEs that are observed with higher frequency and for AESIs (including CRS and ICANS).
Clinical laboratory data | 36 months.
  Clinical laboratory data will be classified by grade according to NCI CTCAE version 5.0 and will be analyzed using summary statistics. The worst on-treatment grades during the treatment period will be summarized.
Overall survival | 36 months
  OS, defined from the date of study registration to the date or death due to any cause.
Patient Frailty | To the time of disease progression.
  Frailty will be measured using the IMWG frailty score and the time for the 4-meter walk test will be recorded.
Frequency and Timing of Hospitalization | 2 weeks.
  Frequency and timing hospitalization will be recorded during the first two weeks of the study treatment.
Patient Quality of Life | To the time of disease progression.
  QoL during treatment measured using the EORTC QOL Questionnaire-C30 instrument EORTC QLQ-C30

OTHER OUTCOMES:
Exploratory outcome BCMA expression (biologic tumor characteristics) | 36 months
  BCMA levels in blood and their relationship to clinical response and progression.
Feasibility, adherence and satisfaction of remote patient monitoring | First 9 days of treatment.
  Feasibility, adherence and satisfaction of remote patient monitoring during the first 9 days of treatment using an outpatient remote monitoring device
Patient satisfaction with the use of the remote monitoring device | First 9 days of treatment.
  Patient satisfaction with the use of the remote monitoring device will be captured using a single, 5-point likert scale question, asked when the device is returned.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Mian, MD, Principal Investigator — McMaster University; Jim Wright, MD, Study Director — OCOG - McMaster University
Locations (4):
- Canada (4):
  - Vancouver Cancer Center, Vancouver, British Columbia
  - Juravinski Cancer Center, Hamilton, Ontario
  - London Health Science Centre - Victoria Hospital, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No